CLINICAL TRIAL: NCT05139095
Title: Camrelizumab Plus Apatinib in Patients With High-risk Gestational Trophoblastic Neoplasia: a Cohort, Open-label, Phase 2 Trial
Brief Title: Camrelizumab Plus Apatinib in Patients With High-risk Gestational Trophoblastic Neoplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GTN-II-001
Record Dates: First submitted 2021-11-06; First posted 2021-12-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-04

CONDITIONS: Gestational Trophoblastic Neoplasia
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Population: ultra high-risk gestational trophoblastic neoplasia
  Interventions: Drug: Camrelizumab plus apatinib CohortA
- Cohort B (Experimental): Population: high-risk chemo-refractory or relapsed gestational trophoblastic neoplasia
  Interventions: Drug: Camrelizumab plus apatinib Cohort B

INTERVENTIONS:
Drug: Camrelizumab plus apatinib CohortA — Camrelizumab (200 mg q2w iv) concomitantly with apatinib (250 mg qd po) and EMA/CO (etoposide, methotrexate, actinomycin D/cyclophosphamide, vincristine, alternate weekly) chemotherapy. For patients with high tumor burden, 1-2 cycles of low-dose chemotherapy will be administered to avoid early death caused by sudden tumor collapse, then followed by standard chemotherapy of EMA/CO. The low-dose chemotherapy will be administered using AE (actinomycin D 500 ug and etoposide 100mg/m2, day 1-3,every 2 week) or EP (etoposide 100 mg/m2 and cisplatin 20 mg/m2, day 1-2, repeated weekly).
  Other Names: Camrelizumab plus apatinib and multi-drug chemotherapy
  Arms: Cohort A
Drug: Camrelizumab plus apatinib Cohort B — Cohort B: Camrelizumab (200 mg q3w iv) concomitantly with apatinib (250 mg qd po) and multi-drug chemotherapy. The multi-drug chemotherapy regimen will be chosen by the investigator (chemotherapy regimen: EMA/CO [etoposide, methotrexate, actinomycin D/cyclophosphamide, vincristine]; or EMA/EP [etoposide, methotrexate and actinomycin-D/etoposide, cisplatin]; or FAEV [floxuridine, actinomycin-D, etoposide, vincristine]). The observation period is 21 days.
  Other Names: Camrelizumab plus apatinib and multi-drug chemotherapy
  Arms: Cohort B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of camrelizumab and apatinib as combination therapy in patients with ultra high-risk (Cohort A) and high-risk chemo-refractory or relapsed (Cohort B) gestational trophoblastic neoplasia (GTN). Eligible patients will receive camrelizumab plus apatinib plus chemotherapy. Treatment will be continued until disease progression, unacceptable toxicity, or withdrawal of consent.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of camrelizumab and apatinib as combination therapy in patients with ultra high-risk (Cohort A) and high-risk chemo-refractory or relapsed (Cohort B) gestational trophoblastic neoplasia (GTN).

Cohort A: Eligible patients will receive camrelizumab (200mg q2w iv) plus apatinib (250 mg qd po) plus chemotherapy. After normalization of serum β-human chorionic gonadotropin (β-hCG) levels, patients will receive 4 cycles of consolidation chemotherapy combined with camrelizumab plus apatinib and then 6 months of camrelizumab plus apatinib as maintenance treatment. Treatment will be continued until completion of treatment, disease progression, unacceptable toxicity, or withdrawal of consent.The primary endpoint is complete remission rate (the proportion of patients achieving complete remission). Secondary endpoints include objective response rate (the proportion of patients achieving complete remission and partial remission), progression-free survival (time from the treatment initiation to disease progression or death, whichever comes first), overall survival (time from the treatment initiation to the date of death or last follow-up), duration of response (time from the first evidence of response to disease progression or death, whichever comes first) and safety.

Cohort B: Eligible patients will receive camrelizumab (200mg q3w iv) plus apatinib (250 mg qd po) plus chemotherapy. Treatment will be continued until disease progression, unacceptable toxicity, or withdrawal of consent. Patients will receive 6 cycles of consolidation therapy if achieving a complete response. The primary endpoint is objective response rate. Secondary endpoints include progression-free survival, duration of response, overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged 18-60 years;
2. Previously untreated patients with ultra high-risk GTN（Cohort A） or high-risk chemo-refractory or relapsed GTN (Cohort B);
3. No previous chemotherapy or radiotherapy for ultra high-risk GTN（Cohort A）and have previously received two or more lines of combination chemotherapies for high-risk chemo-refractory or relapsed GTN (Cohort B);
4. Patients with ultra high-risk GTN (FIGO stages I-III: score ≥13 and stage IV) according to the International Federation of Gynecology and Obstetrics (FIGO) 2000 staging and risk factor scoring system（Cohort A）and patients with a prognostic score ≥7 (Cohort B);
5. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
6. Patients with abnormal serum hCG level (≥5 IU/L);
7. Expected survival ≥ 4 months;
8. The function of vital organs meets the following requirements:

   hemoglobin ≥90 g/L, absolute neutrophil count ≥1·5×109/L, platelets ≥100×109/L; creatinine ≤1·5 × upper limit of normal (ULN), urea nitrogen ≤2·5×ULN; total bilirubin ≤ULN, alanine aminotransferase and aspartate aminotransferase ≤2·5×ULN, albumin ≥25 g/L; thyroid stimulating hormone ≤ULN (if thyroid stimulating hormone is abnormal, normal T3 and T4 can also be acceptable).
9. Female patients of childbearing age must exclude pregnancy and are willing to use a medically approved high-efficiency contraceptive (e.g., intrauterine device, contraceptive or condom) during the study period and within 6 months of the last study drug administration.
10. The patient should be aware of the purpose of the study and the operations required by the study and volunteer to participate in the study before sign the informed consent form.

Exclusion Criteria:

1. Previous treatment with immunotherapy drugs (including antibodies targeting PD-1, PD-L1, cytotoxic T-lymphocyte-associated protein 4, T-cell receptor, chimeric antigen receptor T-cell therapy, and other immunotherapy), anti-angiogenic small-molecule tyrosine kinase inhibitors (such as pazopanib, sorafenib, or regorafenib), or anti-angiogenic monoclonal antibodies (such as bevacizumab); live vaccines injected within 4 weeks before the first dose of study drug; other clinical trials of antitumour drugs within 4 weeks before the first dose of study drug;
2. Other malignancies in the past 3 years;
3. Immunosuppressive drugs used within 14 days prior to the first dose of camrelizumab; any active autoimmune disease or a history of autoimmune disease;
4. Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite with the optimal drug therapy);
5. Grade II or higher myocardial ischemia, myocardial infarction or poorly controlled arrhythmia (females with QTc interval ≥470 ms); grade III to IV cardiac insufficiency according to New York Heart Association (NYHA) criteria, or cardiac color Doppler ultrasound evidence of left ventricular ejection fraction <50%; myocardial infarction, NYHA grade II or above heart failure, uncontrolled angina, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or electrocardiogram suggesting acute ischemia or abnormal active conduction system occurring within 6 months before enrolment;
6. Abnormal coagulation (international normalised ratio >1·5×ULN or prothrombin time >ULN+4 seconds or activated partial thromboplastin time >1·5×ULN), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy;
7. Severe infections within 4 weeks prior to the first dose of study drug (e.g., need of intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever (>38·5°C) during screening or the first dose of study drug;
8. With a history of psychotropic drug abuse and are unable to withdraw the psychotropic drug, or have mental disorders;
9. Major surgery performed within 4 weeks before the first dose of study drug, or open wounds or fractures;
10. Obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction, or sinus or perforation of empty organs within 6 months;
11. Routine urine test indicating urinary protein ++ or more, or confirmed urinary protein ≥1·0 g within 24 hours;
12. Human immunodeficiency virus infection or known acquired immunodeficiency syndrome, active hepatitis B (HBV DNA >500 IU/mL), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the lower limit of the analysis method) or co-infection with hepatitis B and hepatitis C;
13. Other reasons as judged by the investigator.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Complete remission rate | up to one year
  The proportion of patients achieving complete remission. Complete remission is defined as normal serum β-hCG level measured for 3 consecutive weeks.
Cohort B: Objective response rate | up to one year
  The proportion of patients with complete or partial response according to serum β-hCG level. Partial response is defined as a ≥50% decrease in β-hCG level from baseline after 2 cycles.

SECONDARY OUTCOMES:
Cohort A: Objective response rate | up to one year
  The proportion of patients with complete or partial response according to serum β-hCG level.
Cohort A: Progression-free survival | up to one year
  The time from the treatment initiation to disease progression or death, whichever comes first. Disease progression is defined as any increase in serum β-hCG level from baseline after 2 cycles of treatment or the presence of new metastatic lesions.
Cohort A: Overall survival | up to one year
  The time from the treatment initiation to the date of death or last follow-up.
Cohort A: Duration of response | up to one year
  The time from the first evidence of response to disease progression or death, whichever comes first.
Cohort A: Frequency and severity of adverse events | up to one year
  Determine frequency and severity of adverse events as assessed by NCI CTCAE (Version 5.0) which is used to evaluate the grade of adverse events, to observe any adverse event and serious adverse event that occurred in all patients during the clinical study period, including abnormal laboratory examination results, clinical manifestations and vital signs, to record their clinical manifestation characteristics, severity, occurrence time, duration, corresponding treatment and prognosis, and to determine their relationship with the study drug.
Cohort B: Progression-free survival | up to one year
  The time from the treatment initiation to disease progression or death, whichever comes first.
Cohort B: Duration of response | up to one year
  The time from the first evidence of response to disease progression or death, whichever comes first.
Cohort B: Overall survival | up to one year
  The time from the treatment initiation to the date of death or last follow-up.
Cohort B: Frequency and severity of adverse events | up to one year
  Determine frequency and severity of adverse events as assessed by NCI CTCAE (Version 5.0) .

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No